CLINICAL TRIAL: NCT02414893
Title: Hunger/Satiety's Physiopathologic Study in Morbidly Obese Patients: Relation Between Hunger/Satiety, Gastric Emptying, Gallbladder Motility and Peripheral Neurohormonal Signs
Brief Title: Hunger/Satiety's Physiopathologic Study in Morbidly Obese Patients
Status: Completed | Type: Observational
Sponsor: Consorci Sanitari del Maresme (Other)
Responsible Party: Sponsor
Other Study IDs: 15/08
Record Dates: First submitted 2015-03-25; First posted 2015-04-13 (Estimated); Last update posted 2015-04-13 (Estimated); Status verified 2015-04

CONDITIONS: Morbid Obesity
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Non obese
- Morbidly obese
- Sleeve gastrectomy
  Interventions: Procedure: Sleeve gastrectomy

INTERVENTIONS:
Procedure: Sleeve gastrectomy — Laparoscopic vertical gastrectomy as a bariatric procedure.
  Groups: Sleeve gastrectomy

SUMMARY:
The mechanisms that regulate appetite in the morbidly obese are multifactorial and not well-known. Different peripheral signals (such as ghrelin or cholecystokinin) play an important role in the central regulation of appetite and hunger. Postprandial ghrelin and cholecystokinin (CCK) response has also an effect on gastric emptying that, in turn, has an effect on satiety sensation.

On the other hand, bariatric surgery is supposed to affect hunger and satiety in and also promotes changes in gastric emptying which are not clearly defined.

Aim: To better understand the physiologic mechanisms involved in the regulation of hunger and satiety in morbidly obese individuals, especially those related with gallbladder and gastric emptying, as well as those related with the response of the gastrointestinal hormones ghrelin, CCK and glucagon-like peptide-1 (GLP-1), before and after bariatric surgery (sleeve gastrectomy). Methodology: Three groups of individuals will be studied and compared: group A) non obese healthy subjects, group B) morbidly obese subjects and group C) morbidly obese subjects who had had a previous sleeve gastrectomy. In all subjects a standard meal test after a fasting night will be administered and appetite, satiety and hormonal response (ghrelin, CCK, GLP-1 and insulin) during 4 hours post-ingestion assessed, as well as postprandial gallbladder and gastric emptying by means of ultrasonography and the paracetamol absorption technique.

ELIGIBILITY:
Inclusion Criteria:

Group A: non obese individuals (Body Mass Index; BMI < 30 Kg/m2) Group B: Fulfilling the National Health Institute (NHI) criteria for bariatric surgery (BMI higher than 40 Kg/m2 or 35 Kg/m2 when related comorbidities) Group C: Previous morbidly obese individuals who had had a sleeve gastrectomy at least 6 months ago.

Exclusion Criteria:

Group A: previous gastric surgery or gallbladder removal. Group B: previous gastric surgery or gallbladder removal. Group C: previous gallbladder removal.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Group A: non obese healthy individuals Group B: morbidly obese individuals Group C: individuals who had had a previous sleeve gastrectomy as a bariatric procedures
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2009-09; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Hunger and satiety assessment by Visual Analogic Scale | 4 hours

SECONDARY OUTCOMES:
Gastric emptying differences between groups measured by paracetamol absorption test | 4 hours
Gallbladder volume differences between groups measured by ultrasonography | 4 hours
Ghrelin level differences between groups | 4 hours
CCK level differences between groups | 4 hours
GLP-1 level differences between groups | 4 hours
Glucose homeostasis differences between groups | 4 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Consorci Sanitari del Maresme, Mataró, Barcelona, Spain

REFERENCES:
- [Derived] Mans E, Serra-Prat M, Palomera E, Sunol X, Clave P. Sleeve gastrectomy effects on hunger, satiation, and gastrointestinal hormone and motility responses after a liquid meal test. Am J Clin Nutr. 2015 Sep;102(3):540-7. doi: 10.3945/ajcn.114.104307. Epub 2015 Jul 22. PMID 26201818